CLINICAL TRIAL: NCT02675361
Title: Effectiveness of a Transition Program to Empower Adolescents With Congenital Heart Disease in the Transition to Adulthood: the STEPSTONES Project
Brief Title: Effectiveness of a Transition Program for Adolescents With Congenital Heart Disease in the Transition to Adulthood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Swedish Heart Lung Foundation (Other); Swedish Children Heart Association (Unknown); The Swedish Research Council (Other Government); Sahlgrenska University Hospital (Other); Skane University Hospital (Other); Norrlands University Hospital (Other); Karolinska University Hospital (Other); Swedish Council for Working Life and Social Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STEPSTONES-ConHD
Record Dates: First submitted 2016-02-02; First posted 2016-02-05 (Estimated); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Congenital Heart Disease
Keywords: Transfer to adult care; Continuity of patient care; Transition program
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intervention group: transition program (Experimental): Participants come from two clinics and will be randomly allocated to this group. Participants will go through a transition program which will last for 2 years. The intervention will be performed by specialist nurses.
  Interventions: Behavioral: Transition program
- Comparison group (No Intervention): Participants allocated to this group will receive usual care, which includes follow-up visits according to the complexity of the congenital heart disease. Usual care can vary across clinics, however, they all include meeting with a nurse and a physician.
  This is established as a comparison group since there is the risk of contamination in this group.
- Control group (No Intervention): Participants in this group will receive usual care. Follow-up visits will depend on the complexity of the disease.
  Five clinis comprise this section of the study and will be part of an longitudinal, observational study, which investigators will use as a control group.

INTERVENTIONS:
Behavioral: Transition program — Participants will be part of a transition program with eight key components: 1. A transition coordinator; 2. Education on congenital heart disease (CHD), treatments, health behavior, dealing with school, friends; 3. Telephone availability; 4. Information about the Grown-Up Congenital Heart Disease (GUCH) program: 5. Guidance of parents; 6. Meeting with peers: 7. A person-centered transition plan; and 8. Transfer to Grown-Up Congenital Heart Disease clinic. The intervention will be implemented by specialized nurses at the outpatient clinic of pediatric cardiology. Overall, 60 to 90 minutes per patient are spent over the 2.5 years.
  Arms: Intervention group: transition program

SUMMARY:
This study is part of a larger research project known as Swedish Transition Effects Project Supporting Teenagers with chrONic mEdical conditionS (STEPSTONES). This project was created to develop and evaluate transition programs in order to support adolescents with chronic conditions in Sweden. While STEPSTONES has a generic nature, the first transition program that will be evaluated targets adolescents with congenital heart disease (ConHD).

This particular study involves a hybrid experimental design, meaning a randomized controlled trial is embedded in a longitudinal, observational study. This type of design will help to test the effectiveness of a transition program in order to empower adolescents with congenital heart disease in the transition to adulthood and check for potential contamination of the comparison group. We will recruit 210 participants: 140 adolescents will be part of the randomized controlled trial (70 in the intervention arm; 70 in the comparison arm), and 70 participants will be assigned to the observational, longitudinal arm of the study, which serves as control group in an intervention-naive center. Over a period of two years, three assessments will be done during which all participants will be asked to answer a set of questionnaires.

The intervention to be tested involves patient empowerment, education on their ConHD, dealing with school, health behaviors required to maintain good health, guidance of parents, a person-centered transition plan, among others. The study hypothesis is that adolescents with ConHD who received a structured, person-centered transition program over a 2-year period have a higher patient empowerment score than adolescents who receive usual care.

DETAILED DESCRIPTION:
Congenital heart diseases (ConHD) represent 28% of all congenital abnormalities.This population has experienced an increased life expectancy due to improvements in medical services and surgical techniques. Currently, around 90% of them will reach adulthood. Due to the complexity of these disorders, children with ConHD have to be under continuing follow-up. However, when they reach 18 years, they will be transferred to adult care. In order to help the adolescent in the transitions to adulthood and adult care, transitions programs have been proposed as a complex intervention with the objective of maximizing lifelong functioning and potential through appropriate healthcare services.

Patient empowerment is recognized as an essential element of transition interventions.Through the promotion of patient empowerment the adolescents can become active partners in their care and have the knowledge and capacity to make decisions that affect their life and health status.

While the importance of transition programs has been mentioned previously, high level evidence on the effectiveness of these interventions is limited. The purpose of this study is to assess the effectiveness of a transition program for adolescents with congenital heart disease. In order to asses the effectiveness of the transition program the investigators proposed a hybrid experimental design where a randomized controlled trial is embedded in a longitudinal, observational study.

During the course of the study, participants will be part of a transition program or receive usual care before being transferred to adult care. The primary outcome is level of empowerment and secondary outcomes include patient-reported health, illness perception, quality of life, health behaviors, knowledge on congenital heart disease, transition readiness, parental uncertainty and parenting.

The investigators will assess the effectiveness of the transition program by comparing the level of empowerment between the participants who received usual care and those who participated in the transition program. A higher level of empowerment from the group part of the intervention it's expected.

A process and economic evaluation of the intervention will also be undertaken. The process evaluation will evaluate the process of care delivery within the transition program. This information will helped describe the mechanism of impact, explore potential expansion to other chronic conditions and to prepare permanent implementation of the transition program in Sweden.

The economic evaluation entails an impact budget assessment and a cost-effectiveness analysis.

ELIGIBILITY:
Inclusion Criteria:

* Literate
* Swedish-speaking
* Diagnosed with a congenital heart disease
* Age: 16 years

Exclusion Criteria:

* Syndromes affecting cognitive abilities
* Acquired heart diseases
* Heart transplantation

Ages: 16 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 189 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Level of empowerment | Three measurements over a 2-year period.
  Gothenburg Young Persons Empowerment Scale (GYPES) will be used to assess the level of empowerment. This scale was developed by the researchers involved in this study and has been tested in a previous cross sectional study in order to determine its psychometric properties in adolescents with congenital heart disease. The investigators will compare the level of empowerment between groups before and after the transfer of care. Empowerment level will be measured at three different points, when the participants are 16 (baseline), 17 (midterm) and 18 years old (after transfer).

SECONDARY OUTCOMES:
Transition readiness | Three measurements over a 2-year period.
  Readiness for transition questionnaire (adolescent version)
Knowledge | Three measurements over a 2-year period.
  Knowledge scale for adults with congenital malformed hearts
Health behavior | Three measurements over a 2-year period.
  Health behavior scale-congenital heart disease
Patient reported health I | Three measurements over a 2-year period.
  Questionnaire (PedsQL 4.0) (generic and cardiac module)
Quality of life | Three measurements over a 2-year period.
  Linear analog scale
Patient reported health II | Three measurements over a 2-year period.
  Questionnaire (EQ-5D-3L)
Healthcare utilization | Three measurements over a 2-year period.
  Healthcare utilization questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Philip Moons, Principal Investigator — University of Gothenburg and KU Leuven
Locations (7):
- Sweden (7):
  - Children's Heart Center, Queen Silvia Children and Youth Hospital, Gothenburg
  - Children Outpatient Clinic, Linköping University Hospital, Linköping
  - Children's Heart Center, Skåne University Hospital, Lund
  - Child and Adolescent Clinic, Örebro University Hospital, Örebro
  - Children's Outpatient Cardiology Clinic, Astrid Lindgrens Children's Hospital, Stockholm
  - Children's Outpatient Cardiology Clinic, Norrland University Hospital, Umeå
  - Children's Outpatient Cardiology Clinic, Academic Children's Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
Coded files will be available only for research purposes. Information will be given after a letter with the intention of the study has been submitted to the Steering Committee who will determine whether to approve or deny the application.

REFERENCES:
- [Background] Hilderson D, Moons P, Van der Elst K, Luyckx K, Wouters C, Westhovens R. The clinical impact of a brief transition programme for young people with juvenile idiopathic arthritis: results of the DON'T RETARD project. Rheumatology (Oxford). 2016 Jan;55(1):133-42. doi: 10.1093/rheumatology/kev284. Epub 2015 Aug 28. PMID 26320142
- [Background] Hilderson D, Westhovens R, Wouters C, Van der Elst K, Goossens E, Moons P. Rationale, design and baseline data of a mixed methods study examining the clinical impact of a brief transition programme for young people with juvenile idiopathic arthritis: the DON'T RETARD project. BMJ Open. 2013 Dec 2;3(12):e003591. doi: 10.1136/bmjopen-2013-003591. PMID 24302502
- [Background] Knauth Meadows A, Bosco V, Tong E, Fernandes S, Saidi A. Transition and transfer from pediatric to adult care of young adults with complex congenital heart disease. Curr Cardiol Rep. 2009 Jul;11(4):291-7. doi: 10.1007/s11886-009-0042-8. PMID 19563729
- [Background] Moons P, Bovijn L, Budts W, Belmans A, Gewillig M. Temporal trends in survival to adulthood among patients born with congenital heart disease from 1970 to 1992 in Belgium. Circulation. 2010 Nov 30;122(22):2264-72. doi: 10.1161/CIRCULATIONAHA.110.946343. Epub 2010 Nov 22. PMID 21098444
- [Background] McDonagh JE, Kelly DA. The challenges and opportunities for transitional care research. Pediatr Transplant. 2010 Sep 1;14(6):688-700. doi: 10.1111/j.1399-3046.2010.01343.x. Epub 2010 Jun 17. PMID 20557475
- [Background] Small N, Bower P, Chew-Graham CA, Whalley D, Protheroe J. Patient empowerment in long-term conditions: development and preliminary testing of a new measure. BMC Health Serv Res. 2013 Jul 8;13:263. doi: 10.1186/1472-6963-13-263. PMID 23835131
- [Background] Sable C, Foster E, Uzark K, Bjornsen K, Canobbio MM, Connolly HM, Graham TP, Gurvitz MZ, Kovacs A, Meadows AK, Reid GJ, Reiss JG, Rosenbaum KN, Sagerman PJ, Saidi A, Schonberg R, Shah S, Tong E, Williams RG; American Heart Association Congenital Heart Defects Committee of the Council on Cardiovascular Disease in the Young, Council on Cardiovascular Nursing, Council on Clinical Cardiology, and Council on Peripheral Vascular Disease. Best practices in managing transition to adulthood for adolescents with congenital heart disease: the transition process and medical and psychosocial issues: a scientific statement from the American Heart Association. Circulation. 2011 Apr 5;123(13):1454-85. doi: 10.1161/CIR.0b013e3182107c56. Epub 2011 Feb 28. No abstract available. PMID 21357825
- [Derived] Lalji R, Koh L, Francis A, Khalid R, Guha C, Johnson DW, Wong G. Patient navigator programmes for children and adolescents with chronic diseases. Cochrane Database Syst Rev. 2024 Oct 9;10(10):CD014688. doi: 10.1002/14651858.CD014688.pub2. PMID 39382077
- [Derived] Bratt EL, Mora MA, Sparud-Lundin C, Saarijarvi M, Burstrom A, Skogby S, Fernlund E, Fadl S, Rydberg A, Hanseus K, Kazamia K, Moons P. Effectiveness of the STEPSTONES Transition Program for Adolescents With Congenital Heart Disease-A Randomized Controlled Trial. J Adolesc Health. 2023 Oct;73(4):655-663. doi: 10.1016/j.jadohealth.2023.02.019. Epub 2023 Apr 8. PMID 37032211
- [Derived] Acuna Mora M, Sparud-Lundin C, Bratt EL, Moons P. Person-centred transition programme to empower adolescents with congenital heart disease in the transition to adulthood: a study protocol for a hybrid randomised controlled trial (STEPSTONES project). BMJ Open. 2017 Apr 17;7(4):e014593. doi: 10.1136/bmjopen-2016-014593. PMID 28420661